CLINICAL TRIAL: NCT06853795
Title: European E-health Tool for the Appropriate (pre)selection for Spinal Cord Stimulation in Patients with Chronic Pain
Brief Title: Prospective Validation Study of an E-health Tool for Patient Selection for SCS
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Dr. Frank Huygen, Prof. Dr., Erasmus Medical Center
Other Study IDs: SCS e-health tool
Record Dates: First submitted 2025-02-19; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Pain, Chronic
Keywords: SCS; e-health tool; patient selection
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic pain patients eligible for spinal cord stimulation: Patients with chronic pain with a positive decision on SCS. Those receiving either a direct implant or a positive screening trial will be followed at 6 and 12 months after receiving SCS

SUMMARY:
The goal of this observational study is to learn more about the selection of patients with chronic pain for spinal cord stimulation. The main question it aims to answer is to assess the predictive value of an e-health tool for patient outcomes.

Participants will be treated as normal and will be asked to complete patient questionnaires to evaluate their pain relief after receiving spinal cord stimulation. The e-health tool will not be used during the conduct of the study, as patient outcomes will only at the end of the study be compared with the recommendations made by the e-health tool.

DETAILED DESCRIPTION:
This is a multicentre study within Europe, prospectively collecting data from patients with a positive decision on SCS, receiving either a direct implant or an SCS screening trial. Data will be collected by implant centres who have not previously used the e-health tool for SCS patient selection (i.e. tool-naïve). Furthermore, participating centres should declare neither to use the tool during the conduct of study nor on patients included in the study population. In addition, participating implant centres should have previous experience in conducting prospective clinical trials.

Baseline data should be collected at the moment of the final decision on SCS (i.e., after multidisciplinary team consultation if applicable) using an online data capture program:

* General baseline data
* e-Health tool variables
* Centre decision on SCS (direct implant or trial)

Only for patients receiving SCS (direct implant or positive trial), follow-up data at 6 and 12 months will be collected.

Afterwards, the prospectively collected data will be applied to the e-health tool and its recommendations compared with the centre decisions, trial results and patient outcomes.

ELIGIBILITY:
Inclusion criteria

* Age ≥18 years
* Chronic pain with a duration of least 6 months
* One of the following primary indications: Persistent Spinal Pain Syndrome (PSPS) (type 1 and type 2), Complex Regional Pain Syndrome, Neuropathic Pain Syndrome, Ischaemic Pain Syndrome
* Pain severity at least moderate (VAS ≥ 5, on average over the last month) having a substantial impact on daily functioning and quality of life at the discretion of the attending physician
* Insufficiently responding to appropriate trials of medication, conservative management (e.g. physiotherapy) and/or minimally invasive treatments (such as local anaesthetic nerve blocks), and/or experiencing intolerable side effects of these treatments
* No clear benefits of surgery expected

Exclusion criteria

* Unwilling to have an implant
* Unable to manage the device
* Absolute contra-indications for active treatment (e.g. unfit for undergoing SCS, pregnancy, spine- or skin-related infections, coagulation disorder)
* Uncontrolled disruptive psychological or psychiatric disorder at the discretion of the attending physician
* Ongoing alcohol and drug misuse
* Widespread pain
* Lack of reimbursement of SCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain being eligible for spinal cord stimulation and receiving a direct implant or SCS screening trial
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
e-health tool predictive value | 12 months
  Assessment of the predictive value of the panel recommendations (i.e., not recommended, recommended, highly recommended) embedded in the SCS e-health tool for patient outcomes (a). trial outcome: positive/negative, based on Numeric Pain Rating Scale, range 0-10; b).pain-related outcomes after SCS implant: EQ-5D-5L (range 5-25), Brief Pain Inventory (range 0-10), Global Perceived Effect (range 1-7).

SECONDARY OUTCOMES:
Relationship between panel recommendations with centre decisions | 1 week
  Assessment of the relationship between the panel recommendations (i.e., not recommended, recommended, highly recommended) embedded in the SCS e-health tool with the centre decisions (positive=proceed with SCS; negative=no SCS; defer=reassess in a later phase).
Trial results | 1 week
  Assessment of the predictive value of the panel recommendations (i.e., not recommended, recommended, highly recommended) embedded in the e-health tool for trial results (% pain reduction on Numeric Pain Rating Scale; range 0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Herman Stoevelaar, PhD, Study Director — Ismar Healthcare

IPD SHARING:
Plan to Share IPD: No
No data will be shared with researchers not part of the study